CLINICAL TRIAL: NCT03224663
Title: Module Based Learning and Mobile Application Based Learning Regarding Facility Based Newborn Care Among Nursing Students
Brief Title: Effectiveness of Module Based Learning and Mobile Application Based Learning Regarding Facility Based Newborn Care Among Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Minal Kumari, Student, M.Sc Nursing, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 779
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Mobile Application Based Learning
Keywords: Effectiveness; Module based learning; Mobile application based learning; Facility based newborn care; Knowledge; Practices; Nursing students

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Module based learning (Experimental): Module based learning is self-reading method using learner's guide module on FBNC provided by Department of Pediatrics
  Interventions: Other: Module based learning
- Mobile application based learning (Experimental): Mobile application based learning is learning method using android based mobile application on Facility Based Newborn Care provided by Division of Department of Pediatrics "WHO-CC AIIMS FBNC" deals with posters, videos, Modules.
  Interventions: Other: Mobile application based learning

INTERVENTIONS:
Other: Module based learning — self-reading method using learner's guide module on FBNC provided by Department of Pediatrics.administered 45 minutes
  Arms: Module based learning
Other: Mobile application based learning — learning method using android based mobile application on Facility Based Newborn Care provided by Division of Department of Pediatrics "WHO-CC AIIMS FBNC" deals with posters , videos , Modules.administered 45 minutes
  Arms: Mobile application based learning

SUMMARY:
The study evaluates the effectiveness of Module based learning and Mobile application based learning regarding Facility based newborn care among nursing students.Total 70 Nursing students were randomly allocated to MBL and MABL group . First 35 students received MBL based teaching and next 35 students received MABL teaching.

DETAILED DESCRIPTION:
a comparative study was done to assess the effectiveness of Module based learning and Mobile application based learning regarding Facility based newborn care among nursing students.

MODULE GROUP

Day 1: Pre assessment of Knowledge through Structured knowledge questionnaire was done and practice through observation checklist by OSCE method .

Day 2: Module based Teaching administered to nursing students who were present on the data collection. Teaching and Hands on sessions were given to students by investigator. Introduction regarding Module and topics: Prevention of infection (Hand washing), Kangaroo Mother Care, Feeding of normal and low birth weight babies (Attachment during feeding, Paladai Feeding), Common Procedures (Oxygen administration, Insertion and Orogastric Tube Feeding, Weight Recording of a Newborn)

Day 15th = Post-test of Knowledge through Structured knowledge questionnaire was done in BSc. Nursing 3rd year classroom and practice through observation checklist by OSCE method Post-test of knowledge took 45 minutes.

MOBILE APPLICATION BASED GROUP

Day 16th = Pre assessment of Knowledge through Structured knowledge questionnaire was done in BSc. Nursing 3rd year classroom of M.M Institute of Nursing and practice through observation checklist by OSCE method

Day 17th = Mobile Application based Teaching administered to nursing students who were randomly selected. Teaching and videos were given to students by investigator in MM Institute of Nursing.

Introduction regarding Mobile Application and topics: Modules on Normal baby, At Risk baby, Sick Newborn, Videos on Attachment during feeding, Paladai Feeding, Oxygen administration, Kangaroo Mother Care, Insertion and Orogastric Tube Feeding, Weight Recording of a Newborn, Hand washing, Posters on Hand washing, Kangaroo Mother Care

Day 30th = Post-assessment of Knowledge through Structured knowledge questionnaire was done and practice through OSCE method

ELIGIBILITY:
Inclusion Criteria:

* BSc Nursing 3rd. Year students who were present at the time of data collection

Exclusion Criteria:

* BSc Nursing 3rd. Year students who were not having Android phone in MABL group

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Knowledge scores measured by structured knowledge questionnaire | 45 minutes
  the ability of nursing students to respond correctly to questions regarding FBNC as evidenced by knowledge scores measured by structured knowledge questionnaire and categorized as Very Good (≥80%), Good (65-79%), Average (51-64%) and Below Average (≤50%).

CONTACTS AND LOCATIONS:
Overall Officials: Minal Kumari, M.Sc. Nursing, Principal Investigator — Maharishi Markandeshwar University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franko OI, Tirrell TF. Smartphone app use among medical providers in ACGME training programs. J Med Syst. 2012 Oct;36(5):3135-9. doi: 10.1007/s10916-011-9798-7. Epub 2011 Nov 4. PMID 22052129
- [Background] Thukral A, Joshi M, Joshi P, Prakash V, Adkoli BV, Deorari AK. Apps for management of sick newborn: evaluation of impact on health care professionals. J Trop Pediatr. 2014 Oct;60(5):370-6. doi: 10.1093/tropej/fmu032. Epub 2014 Jun 12. PMID 24924579